CLINICAL TRIAL: NCT06231199
Title: Combined Effect of Foam Roller and Gastrocnemius Release on Plantar Fasciitis
Acronym: MTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Samir Mohamed Bagory, principle investigator: aya samir mohamed bagory, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004276
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Plantar Fascitis
Keywords: foam roller; gastrocnemius release; plantar fascitis

STUDY DESIGN:
Intervention Model Description: foam roller combined with gastrocnemius release and conventional treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gastrocnemius release (Experimental): the patients will receive gastrocnemius release manually and by foam roller three times a week for four weeks plus conventional treatment
  Interventions: Other: gastrocnemius release; Other: conventional treatment
- conventional treatment (Active Comparator): the patients will receive conventional treatment three times a week for four weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: gastrocnemius release — The patient will be prone to lying and the therapist will stand at the side of the patient's leg. The therapist uses both hands in cross-hand pattern (Figure 10a and 10b). Myofascial Release will be performed for 20 repetitions, then gastrocnemius release by foam roller;This involved long sitting, with the affected leg will be extended on the foam roller and foot relaxed. The non-affected leg will be flexed at knee so that the foot will be rested on the floor. The participants will be instructed to use their arms and non_affected foot to propel their body back and forth from the popliteal fossa to Achilles tendon in continuous motion. then patients perform plantar fascia realise from standing by foam roller
  Arms: gastrocnemius release
Other: conventional treatment — the patients will receive conventional treatment in the form of ultrasound therapy (continuous mode/1MHZ) followed by plantar fascia stretch and inctruction

SUMMARY:
this study will be conducted to investigate the efficacy of combining foam roller and gastrocnemius release on pain intensity level, dorsi flexion range of motion of ankle joint ,dorsi flexion range of motion of big toe and foot function in subjects with plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis refers to degeneration and inflammation of the proximal plantar fascia. The condition presents with plantar medial heel pain, often exacerbated following periods of inactivity, such as upon waking in the morning.The term "plantar fasciitis" has been quoted for years, but this is a misnomer as inflammatory cells are not present in biopsies from involved fascia. Therefore, advocate the terminology "plantar fasciitis" to explain the syndrome characterized by pain along the proximal plantar fascia and its attachment in the area of the calcaneal tuberosity with function impairment, implying a more chronic degenerative process than acute heel pain.Research found that both stretching and foam rolling techniques helped reduce pain and increase the ROM. However, the effectiveness of foam rolling was superior to stretching in terms of increased pressure pain thresholds (PPTs) at gastrocnemius and soleus. there was a gap in the previous literature in combined effect of gastrocnemius release and foam roller in managing plantar fasciitis and assessing dorsi flexion range of motion of both big toe and ankle joint along with pain assessment and foot function. sixty patients with planter fascitis will be assigned randomly to two groups; first one will receive manual and foam roller release of gastrocnemius and conventional treatment and the other one will receive conventional treatment only.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 years and 60 years
* heel pain in the morning with first step, insidious sharp pain under the heel, tenderness on medial calcaneus and symptoms decreasing with slight activity (like walking) and worsening toward the end of the day

Exclusion Criteria:

* Infective conditions of foot, tumor, calcaneal fracture
* Metal implant around ankle
* Dermatitis, acute sepsis and anesthetic areas
* Subject with impaired circulation to lower extremities
* Subject with referred pain due to sciatica
* Corticosteroids
* Injection in heel preceding 3 month
* Patient who cannot co-operate
* history of flat foot

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-04-25 (Estimated)

PRIMARY OUTCOMES:
pain intensity level | up to four weeks
  visual analogue scale will be used for assess pain intensity level. VAS was a 10-cm-long horizontal line with no pain and worst possible pain at the extremes of the line
ankle dorsiflexion | up to four weeks
  Electro goniometers are electronic versions of the standard goniometers used in the clinic to measure ankle dorsiflexion ROM
foot function | up to four weeks
  The foot function index (questionnaire) will be used to assess foot function. it consists of 23 self-reported items divided into 3 subcategories based on patient values: pain, disability and activity limitation. The patient has to score each question on a scale from 0 (no pain or difficulty) to 10 (worst pain imaginable or so difficult it requires help)

SECONDARY OUTCOMES:
big toe range of motion | up to four weeks
  Electro goniometers are electronic versions of the standard goniometers used in the clinic to measure big toe range of motion